CLINICAL TRIAL: NCT00506831
Title: A Pilot Study of Imatinib in the Treatment of Refractory Systemic Sclerosis
Brief Title: Imatinib in Systemic Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lorinda S Chung, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9598; 9598
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib mesylate (Experimental): 100 mg daily and increase by 100mg daily every 2 weeks to a maximum of 400 mg daily as tolerated
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — 100 mg orally daily increased by 100 mg/day every 2 weeks to maximum of 400 mg daily as tolerated. Treatment for 6 months total.

SUMMARY:
Systemic sclerosis (SSc) is an autoimmune disease characterized by fibrosis of the skin and internal organs and widespread vasculopathy. Patients with SSc are classified according to the extent of cutaneous sclerosis: patients with limited SSc have skin thickening of the face, neck, and distal extremities, while those with diffuse SSc have involvement of the trunk, abdomen, and proximal extremities as well. The disease course varies depending on the subtype of SSc. However, common features that result in significant morbidity and mortality, in addition to cutaneous fibrosis, include Raynaud's phenomenon and digital ulcerations, interstitial lung disease (ILD), and pulmonary arterial hypertension (PAH). Current therapeutic options for patients with SSc and these clinical manifestations have shown limited efficacy.

Imatinib antagonizes specific tyrosine kinases that mediate fibrotic pathways involved in the pathogenesis of SSc, including c-Abl, a downstream mediator of transforming growth factor (TGF)-beta, and platelet derived growth factor (PDGF) receptors. The efficacy of imatinib has also been reported in the treatment of patients with refractory idiopathic PAH through its effects on vascular remodeling. Based on the mechanism of action and preliminary patient data, we hypothesize that imatinib may be effective in the treatment of the fibrotic and vasculopathic features of patients with SSc. This is an open label pilot study to evaluate the safety and efficacy of imatinib in patients with progressive SSc refractory to other treatment(s). Validated measures of skin thickness and disease activity will be determined over 6-months of therapy and compared with baseline measures.

ELIGIBILITY:
Inclusion Criteria:

Adults with refractory diffuse or limited SSc and any or all of the following: Progressive cutaneous fibrosis, Interstitial lung disease, Pulmonary arterial hypertension, Digital ulcerations.

Exclusion Criteria:

Uncontrolled congestive heart failure, hypertension, or coronary artery disease.

HIV, hepatitis B, and/or hepatitis C infection. Serious infection within the past month. Significant hematologic, renal, or hepatic abnormalities. Concurrent use of intravenous immunoglobulin or cyclophosphamide within 4 weeks of the first treatment dose.

Concurrent use of a biologic agent (ie. etanercept, infliximab, adalimumab, abatacept) within 8 weeks of the first treatment dose (6 months for rituximab).

Women who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorinda S Chung, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Whitfield ML, Finlay DR, Murray JI, Troyanskaya OG, Chi JT, Pergamenschikov A, McCalmont TH, Brown PO, Botstein D, Connolly MK. Systemic and cell type-specific gene expression patterns in scleroderma skin. Proc Natl Acad Sci U S A. 2003 Oct 14;100(21):12319-24. doi: 10.1073/pnas.1635114100. Epub 2003 Oct 6. PMID 14530402
- [Result] Chung L, Fiorentino DF, Benbarak MJ, Adler AS, Mariano MM, Paniagua RT, Milano A, Connolly MK, Ratiner BD, Wiskocil RL, Whitfield ML, Chang HY, Robinson WH. Molecular framework for response to imatinib mesylate in systemic sclerosis. Arthritis Rheum. 2009 Feb;60(2):584-91. doi: 10.1002/art.24221. PMID 19180499

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate: All patients were treated with imatinib mesylate at a mean dosage of 300 mg daily.
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 9
Completed | 7
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Modified Rodnan Skin Score at 6 Months Compared to Baseline
Description: Modified Rodnan skin score (mRSS) on scale of 0 (no skin disease) to 51 severe skin disease. %change in mRSS=(score at 6 months - baseline score)/baseline score. Negative values indicate improvement in skin disease. Clinical important improvement defined as > 25% improvement.
Time Frame: 6 months compared to baseline
Population: Participants who completed the protocol were included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of change in MRSS
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 7
percentage of change in MRSS | -32 (22)
Statistical Analysis 1: Comparison: Imatinib Mesylate; Null hypothesis is that the mRSS is not significantly different at month 6 compared with baseline. Paired t-test was used to compare the mean mRSS at month 6 compared with baseline; Test type: Superiority or Other; p = 0.005, t-test, 2 sided

2. Secondary Outcome: Change in Pulmonary Function Tests at 6 Months Compared to Baseline
Description: Change in % predicted Forced Vital Capacity (FVC) at 6 months compared to baseline. FVC is the volume of air that can forcibly be blown out after taking a full breath. FVC% predicted is defined as FVC% of the patient divided by the average FVC% in the population for any person of similar age, sex and body composition.
Time Frame: 6 months compared to baseline
Population: Participants with available data were included in the analysis
Measure: Mean (Full Range); unit: FVC% predicted
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 5
FVC% predicted | 0 [-7 to 10]

3. Secondary Outcome: Change in Digital Ulcerations at 6 Months Compared to Baseline
Description: Number of digital ulcers as measured by physician assessment at 6 months compared to baseline
Time Frame: 6 months compared to baseline
Population: No data were collected for this outcome measure
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Scleroderma Health Assessment Questionnaire at 6 Months Compared to Baseline
Description: Change in Health Assessment Questionnaire disability index at 6 months compared to baseline. The Questionnaire is comprised of a 20 question instrument pertaining to specific activities with possible integer responses of 0 (without any difficulty) to 3 (unable to do), and five additional scleroderma-specific visual analog scale (VAS) domains with possible values ranging from 0.0 to 15.0. The 20 questions are divided into eight domains. A mean score is calculated for each domain ranging from 0 to 3. A composite score is calculated by dividing the summed domain scores by the number of domains answered. The composite score is reported, falling between 0 and 3 on an ordinal scale. The scores are interpreted as 0 (no impairment in function) to 3 (maximal impairment of function).
Time Frame: 6 months compared to baseline
Population: Participants with available data were included in the analysis
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 5
units on a scale | -.35 [-.88 to .38]

5. Secondary Outcome: Change in Dermal Thickness and Collagen Separation on Cutaneous Histopathology at 6 Months Compared to Baseline
Time Frame: 6 months compared to baseline
Population: Participants with available data were included in the analysis
Measure: Number; unit: mm
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 1
mm | -.5

6. Secondary Outcome: Change in Serum Cytokine Profile at 6 Months Compared to Baseline
Time Frame: 6 months compared to baseline
Population: No data were collected for this outcome measure
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

7. Secondary Outcome: Cell Types That Contribute to the Gene Expression Changes Associated With Imatinib Therapy
Description: To determine which cell types may be contributing to the gene expression changes associated with imatinib therapy, imatinib-responsive genes were isolated from from patient biopsies. From the total number of imatinib-responsive genes that were isolated, the percentage that came from endothelial cells, fibroblasts, B-cells, and multiple cell types was calculated. Reported values do not total to 100% because of rounding.
Time Frame: 6 months compared to baseline
Population: Participants with available data were included in the analysis
Measure: Number; unit: percentage of isolated genes
Units Other Than Participants: Isolated imantinib-responsive genes
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 2
Number analyzed (Isolated imantinib-responsive genes) | 1050
percentage of isolated genes
  Endothelial cells | 13
  Fibroblasts | 26
  B-cells | 8
  Multiple cell types | 52

8. Secondary Outcome: Change in Serum Autoantibody Profile at 6 Months Compared to Baseline
Time Frame: 6 months compared to baseline
Population: No data were collected for this outcome measure
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=9)
Death (Infections and infestations) | 1 (1) — Patient experienced pneumonia, was found to be neutropenic, and died of sepsis prior to week 8 assessment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=9)
infection (Infections and infestations) | 7 (11) — 7 patients (78%) experienced infections throughout study:
edema (Blood and lymphatic system disorders) | 6 (6)
gastrointestinal symptoms (Gastrointestinal disorders) | 6 (10)
new digital ulcers (Vascular disorders) | 2 (2)
fever (Infections and infestations) | 1 (1)
neutropenia (Immune system disorders) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1)
hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
oral ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
blurry vision (Eye disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
hypokalemia (Renal and urinary disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
keratitis (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open label, uncontrolled study. Small study population at a single center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No